CLINICAL TRIAL: NCT05690711
Title: Efficacy and Safety of Intravenous HRS8179 on Brain Swelling After Large Hemispheric Infarction: a Randomised, Double-blind, Placebo-controlled Phase II Trial
Brief Title: A Trial of HRS8179 on Brain Swelling After Large Hemispheric Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS8179-201
Record Dates: First submitted 2022-12-27; First posted 2023-01-19 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-05

CONDITIONS: Brain Swelling, Large Hemispheric Infarction
MeSH Terms: conditions — Brain Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS8179 (Experimental)
  Interventions: Drug: HRS8179
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS8179 — HRS8179 injection
  Arms: HRS8179
Drug: Placebo — physiological saline
  Arms: Placebo

SUMMARY:
The primary objective is to explore if HRS8179 could improve midline shift at 72 hours (or at time of decompressive craniectomy or comfort measures only, if earlier) in participants with large hemispheric infarction. The secondary objective is to explore if HRS8179 could improve acute neurologic status, functional outcomes, treatment requirements and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and voluntarily participate in this research, and sign the informed consent form (the informed consent form can be signed voluntarily by the person or legal representative);
2. Aged 18~80, regardless of gender;
3. A clinical diagnosis of acute ischemic stroke in the middle cerebral artery (MCA) territory;
4. NIHSS ≥ 10 points at screening;
5. A large hemispheric infarction is defined as: lesion volume of 80 to 300 cm3 on magnetic resonance imaging (MRI) diffusion-weighted imaging (DWI), or computed tomography perfusion (CTP).
6. The study drug initiated must be no later than 10 hours when stroke onset;

Exclusion Criteria:

1. The investigator judges that the subject may withdrawn the supportive treatment on the first day; The investigator believes that there is evidence indicating a concurrent infarction in the contralateral hemisphere sufficiently serious to affect functional outcome.3. There are clinical signs of brain hernia;
2. CT/MRI suggested that the anterior septal/pineal excursion was >2 mm due to brain edema;
3. CT/MRI indicates cerebral hemorrhage (excluding small ecchymosis/punctate hemorrhage);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
The change between baseline and 72-78 hours in midline shift measured by MRI or CT | Baseline up to 72 hours

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) Score | Day 90
Overall survival | Baseline up to Day 90
Number of Participants Who Achieved mRS 0-4 | Day 90
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided